CLINICAL TRIAL: NCT04590794
Title: A Prospective Observational Study on Assessment of the Soluble Urokinase Plasminogen Activator Receptor in Adult Patients With Covid-19
Brief Title: SuPAR in Adult Patients With Covid-19
Acronym: SPARCOL
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Chalkias, MD, PhD, Asst. Professor of Anesthesiology, University of Thessaly
Other Study IDs: UTHDA-AC03
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Covid19
Keywords: covid 19; organ injury; outcome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid 19: Patients admitted with covid 19
  Interventions: Diagnostic Test: Soluble Urokinase Plasminogen Activator Receptor

INTERVENTIONS:
Diagnostic Test: Soluble Urokinase Plasminogen Activator Receptor — Participants will undergo sampling of peripheral venous blood, immediately after admission. Blood samples drawn from all patients and EDTA plasma will be stored at -80° C until later measurement. Plasma suPAR levels will be determined using the suPARnostic® ELISA assay (ViroGates, Denmark), which is based on a simplified double monoclonal antibody sandwich ELISA assay whereby samples and peroxidase-conjugated anti-suPAR are first mixed together and then incubated in anti-suPAR pre-coated micro wells. The recombinant suPAR standards of the kit are calibrated against healthy human blood donor samples. suPAR concentrations are determined as ng/mL plasma.
  Other Names: suPAR

SUMMARY:
The biomarker soluble urokinase plasminogen activator receptor (suPAR) is the soluble form of the cell membrane-bound protein urokinase plasminogen activator receptor (uPAR), which is expressed mainly on immune cells, endothelial cells, and smooth muscle cells. SPARCOL is a multi-center prospective observational study aiming to investigate if suPAR measured at admission can predict the risk of future complications and mortality in adults patients with Covid-19. The study will include approximately 500 patients and will be one of the largest so far. The study has been registered at Clinical Trials.gov and has been approved by the Institutional Review Board of the University Hospital of Larisa.

Consecutive adult patients (≥ 18 years ) who are admitted to the Hospital due to Covid-19 will be screened for inclusion. Participants will undergo sampling of peripheral venous blood, immediately after admission. Blood samples drawn from all patients and EDTA plasma will be stored at -80° C until later measurement. Plasma suPAR levels will be determined using the suPARnostic® ELISA assay (ViroGates, Denmark).

The primary endpoint will be the presence of respiratory complications, admission to ICU, and survival at 30 days. Secondary endpoints are also included, such as organ injury, hospital length of stay, and survival.

Data analysis will be based on predefined data points on a prospective data collection form.

DETAILED DESCRIPTION:
BACKGROUND

Soluble urokinase plasminogen activator receptor

The biomarker soluble urokinase plasminogen activator receptor (suPAR) is the soluble form of the cell membrane-bound protein urokinase plasminogen activator receptor (uPAR), which is expressed mainly on immune cells, endothelial cells, and smooth muscle cells. uPAR is released during inflammation or immune activation, and therefore the suPAR level reflects the extent of immune activation in the individual. All human beings have a baseline level of suPAR that is individually determined and increases with age. Studies have shown that the suPAR level is associated with morbidity and mortality in a number of acute and chronic diseases and in the general population. The suPAR level is elevated across diseases, and not solely associated with one specific disease. Therefore, suPAR is applicable as a prognostic marker and not as a diagnostic marker. This characteristic may be utilized for risk stratification in unselected patients.

Originally, uPAR was proven a receptor for urokinase (uPA) which splits plasminogen into active plasmin. Moreover, uPAR interacts with other proteins and plays a role in several important cell processes like migration, adhesion, angiogenesis, proliferation, and chemotaxis. The suPAR protein was discovered in 1991, when it was found to be a marker of cancer progression. In recent years, several studies have shown that suPAR is associated with a number of chronic diseases (including cardiovascular, hepatic, renal, and pulmonary diseases), and that the level is a predictor of a negative outcome of various infectious diseases (tuberculosis, HIV, malaria, sepsis, meningitis, pneumonia) and in critically ill patients.

Across diseases, the suPAR level discriminates non-survivors from survivors. suPAR reflects the level of chronic inflammation, and therefore it has been studied as a potential marker of development of diseases, and studies have shown that an elevated level predicts development of chronic diseases and cancer in the general population. The suPAR blood level is stable with no diurnal variation and no changes following fasting, while suPAR can be measured in blood, plasma, urine, cerebrospinal fluid, ascites fluid and pleural fluid. The level increases and decreases with progression and improvement of a disease, respectively, but more slowly compared to e.g. C-reactive protein (CRP). The normal suPAR plasma level is 2-3 ng/mL in healthy individuals, about 3-4 ng/mL in unselected patients in emergency departments, and about 9-10 ng/mL in critically ill patients.

suPAR in intensive care

In critically ill patients, the suPAR level is significantly increased. suPAR is an independent prognostic marker, and the change over time correlates with organ dysfunction. suPAR is elevated and has a prognostic value in patients with: SIRS (systemic inflammatory response syndrome), sepsis/septic shock, burn injuries, and traumatic brain injuries. The suPAR level reflects the body's immune response to infections, and the level increases with the severity of the infection. In patients with organ dysfunction, the suPAR value is often a two-digit value. In particular hepatic and renal dysfunction affects the suPAR level. suPAR has been studied in patients with SIRS who were acutely admitted to the emergency department (n=902). The studies showed that suPAR is a stronger marker of 2-day, 30-day, and 90-day mortality than age, CRP, IL-6, creatinine, and procalcitonin. However, for diagnostic purposes, IL-6 and CRP are superior to suPAR in predicting a positive blood culture. A Greek multicenter study including 1914 patients with sepsis showed that suPAR is a strong predictor of mortality, and that a suPAR level above 12 ng/mL is linked to a >80% sensitivity for mortality and a negative predictive value of 94.5%. In addition, the prognostic value of suPAR in patients with sepsis is independent of relevant covariates like APACHE score, CRP, etc.

In patients with burn injuries and inhalation trauma requiring mechanical ventilation, the plasma suPAR level and bronchoalveolar lavage fluid level correlate to IL-6 and coagulation factors. An elevated plasma suPAR level is associated with prolonged Intensive Care Unit (ICU) stay and the duration of mechanical ventilation. The suPAR level is elevated in patients with traumatic brain injury. In trauma patients who suffered a brain injury within 12 hours prior to blood sampling, the mean suPAR level is 14.9 ng/mL ± 6.9 vs. 2.8 ng/mL ± 0.7 in control subjects. In these patients suPAR is associated with severity of the brain injury and with mortality.

suPAR and acute respiratory distress syndrome

Mortality rates of patients with the acute respiratory distress syndrome (ARDS) are high. Biological markers as well as disease severity scoring systems may be useful for risk stratification and the creation of homogenous patient groups in clinical trials. However, currently no single biological marker has been found to have sufficient discriminative value for accurate prediction of mortality or bedside decision making in ARDS patients in the clinical setting The first study that investigated the association between plasma suPAR and mortality in a cohort of ARDS patients was published in 2015. In that study, plasma levels of suPAR were higher with increasing severity of ARDS, and higher in patients who died in the ICU. Furthermore, higher plasma suPAR levels were associated with less ventilator- and ICU-free days.

In a prospective, multicenter, observational study including mechanically ventilated ICU patients, low concentrations of suPAR were predictive for survival and high concentrations for renal replacement therapy and mortality. The authors concluded that SuPAR may be used for screening for patients with potentially good survival, while its association with renal replacement therapy may supply an early warning sign for acute renal failure. Several other authors have evaluated the predictive value of suPAR regarding the risk of ARDS in sepsis patients, and reported a correlation/association with disease severity, inflammation and mortality.

AIM

SPARCOL is a multi-center observational study aiming to investigate if suPAR measured at admission can predict the risk of future complications and mortality in adults patients with Covid-19.

METHODS

Design

This is a prospective observational study designed in accordance with the declaration of Helsinki. The study will be registered at Clinical Trials.gov and has been approved by the Institutional Review Board of the University Hospital of Larisa, under the reference number 17543.The study will be approved by the IRB of each of the participating centers.

Patient eligibility

Inclusion criteria will be: (1) adult (≥18 years old) patients hospitalized primarily for COVID-19; (2) a confirmed SARS-CoV-2 infection diagnosed through reverse transcriptase polymerase chain reaction test of nasopharyngeal or oropharyngeal samples; and (3) at least one blood sample collected at admission and stored for biomarker testing. Patients with confirmed SARS-CoV-2 infection who will not be primarily admitted for COVID-19 and patients with incomplete data will be excluded.

Sampling and laboratory measurements

Participants will undergo sampling of peripheral venous blood, immediately after admission. Blood samples drawn from all patients and EDTA plasma will be stored at -80° C until later measurement. Plasma suPAR levels will be determined using the suPARnostic® ELISA assay (ViroGates, Denmark), which is based on a simplified double monoclonal antibody sandwich ELISA assay whereby samples and peroxidase-conjugated anti-suPAR are first mixed together and then incubated in anti-suPAR pre-coated micro wells. The recombinant suPAR standards of the kit are calibrated against healthy human blood donor samples. suPAR concentrations are determined as ng/mL plasma.

Outcomes

The primary endpoint will be the presence of respiratory complications [need of non-invasive ventilation (CPAP-BiPAP), hi-flow nasal oxygen, or mechanical ventilation], admission to ICU, and survival at 30 days.

Secondary endpoints will be hypotension (defined as systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg for 3 minutes or more), need for vasoactive drugs (need for vasoactive drugs not planned before and/or continuous infusion), and/or acute new cardiovascular disorder (atrial fibrillation, sustained ventricular tachycardia, supraventricular tachycardia, myocardial infarction, pericarditis, myocarditis, cardiogenic shock, and/or cardiac arrest), renal failure, duration of mechanical ventilation, reintubation, hospital length of stay, length of stay in ICU and readmission.

Data Collection and Monitoring

Data analysis will be based on predefined data points on a prospective data collection form. The staff will be blinded to measurements until the end of the study and all data are analyzed. Clinical monitoring throughout the study will be performed to maximize protocol adherence, while an independent Data and Safety Monitoring research staff will monitor safety, ethical, and scientific aspects of the study. Data collection will also include demographics, general blood count, C-reactive protein, APACHE II, and SOFA.

Data management

The goal of the clinical data management plan is to provide high-quality data by adopting standardized procedures to minimize the number of errors and missing data, and consequently, to generate an accurate database for analysis. Remote monitoring will be performed to signal early aberrant patterns, issues with consistency, credibility and other anomalies. Any missing and outlier data values will be individually revised and completed or corrected whenever possible.

Sample size

This study will include approximately 500 patients. Based on international and national epidemiological data, we anticipate that approximately 30% of the included patients will reach the primary endpoints.

Ethics and dissemination

The study will be performed according to national and international guidelines. The study will begin after approval has been obtained from the Hospital's Institutional Review Board, according to local regulation. Prospective written informed consent will be requested before inclusion of all eligible patients based on the Review Board's decision.

Competing interests None declared.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* patients hospitalized primarily for Covid 19
* confirmed SARS-CoV-2 infection diagnosed through RT-PCR test of nasopharyngeal or oropharyngeal samples
* at least one blood sample collected during the hospitalization and stored for biomarker testing

Exclusion Criteria:

* patients with confirmed SARS-CoV-2 infection who will not be primarily admitted for COVID-19
* patients with incomplete data

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients who are admitted to the Hospital due to Covid-19
Sampling Method: Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
respiratory complications | Up to 8 weeks
  need of non-invasive ventilation (CPAP-BiPAP), hi-flow nasal oxygen, or mechanical ventilation

SECONDARY OUTCOMES:
Hypotension | Up to 8 weeks
  systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg for 3 minutes or more
need for vasoactive drugs | Up to 8 weeks
  need for vasoactive drugs not planned before and/or continuous infusion
Number of participants with acute new cardiovascular disorder | Up to 8 weeks
  Number of participants with atrial fibrillation, sustained ventricular tachycardia, supraventricular tachycardia, myocardial infarction, SPARCOL Study April 12, 2020 7 pericarditis, myocarditis, cardiogenic shock, and/or cardiac arrest
Number of participants with organ failure | Up to 8 weeks
  Number of participants with any organ failure
Number of participants with overall survival up to 8 weeks | Up to 8 weeks
  Number of participants who survive up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Chalkias, PhD, Principal Investigator — University of Thessaly
Locations (1):
- University Hospital of Larisa, Department of Anesthesiology, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Chalkias A, Mouzarou A, Samara E, Xanthos T, Ischaki E, Pantazopoulos I. Soluble Urokinase Plasminogen Activator Receptor: A Biomarker for Predicting Complications and Critical Care Admission of COVID-19 Patients. Mol Diagn Ther. 2020 Oct;24(5):517-521. doi: 10.1007/s40291-020-00481-8. PMID 32613288
- [Background] Azam TU, Shadid HR, Blakely P, O'Hayer P, Berlin H, Pan M, Zhao P, Zhao L, Pennathur S, Pop-Busui R, Altintas I, Tingleff J, Stauning MA, Andersen O, Adami ME, Solomonidi N, Tsilika M, Tober-Lau P, Arnaoutoglou E, Keitel V, Tacke F, Chalkias A, Loosen SH, Giamarellos-Bourboulis EJ, Eugen-Olsen J, Reiser J, Hayek SS; International Study of Inflammation in COVID-19. Soluble Urokinase Receptor (SuPAR) in COVID-19-Related AKI. J Am Soc Nephrol. 2020 Nov;31(11):2725-2735. doi: 10.1681/ASN.2020060829. Epub 2020 Sep 22. PMID 32963090
- [Background] Ge H, Wang X, Yuan X, Xiao G, Wang C, Deng T, Yuan Q, Xiao X. The epidemiology and clinical information about COVID-19. Eur J Clin Microbiol Infect Dis. 2020 Jun;39(6):1011-1019. doi: 10.1007/s10096-020-03874-z. Epub 2020 Apr 14. PMID 32291542